CLINICAL TRIAL: NCT05705401
Title: A Phase III Randomized Trial of Radiotherapy Optimization for Low-Risk HER2-Positive Breast Cancer (HERO)
Brief Title: Testing Radiation and HER2-targeted Therapy Versus HER2-targeted Therapy Alone for Low-risk HER2-positive Breast Cancer
Acronym: HERO
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: NRG Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Alliance for Clinical Trials in Oncology (Other); Eastern Cooperative Oncology Group (Network); SWOG Cancer Research Network (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NRG-BR008; 5U10CA180868 (NIH); NCI-2022-09157 (Other: NCI)
Record Dates: First submitted 2023-01-05; First posted 2023-01-30 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-08

CONDITIONS: HER2-positive Breast Cancer

STUDY DESIGN:
Intervention Model Description: Subjects who are receiving standard of care systemic HER2-targeted therapies are randomized to standard of care adjuvant breast radiation or no breast radiation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care Adjuvant Breast Radiation (Active Comparator): Patients continue to receive their current planned adjuvant breast radiation and systemic HER2-targeted therapies
  Interventions: Radiation: Standard of Care Adjuvant Breast Radiation
- Standard of Care HER2-targeted Therapy Without Adjuvant Breast Radiation (Active Comparator): Patients continue to receive their current systemic HER2-targeted therapy without breast adjuvant radiation
  Interventions: Drug: Standard of Care HER2-targeted Therapy Without Adjuvant Breast Radiation

INTERVENTIONS:
Radiation: Standard of Care Adjuvant Breast Radiation — adjuvant breast radiotherapy per the current standard of care
  Arms: Standard of Care Adjuvant Breast Radiation
Drug: Standard of Care HER2-targeted Therapy Without Adjuvant Breast Radiation — participants are randomized to continue their standard of care systemic HER2-targeted therapy without adjuvant breast radiotherapy
  Arms: Standard of Care HER2-targeted Therapy Without Adjuvant Breast Radiation

SUMMARY:
This Phase III trial compares the recurrence-free interval (RFI) among patients with early-stage, low risk HER2+ breast cancer who undergo breast conserving surgery and receive HER2-directed therapy, and are randomized to not receive adjuvant breast radiotherapy versus those who are randomized to receive adjuvant radiotherapy per the standard of care.

DETAILED DESCRIPTION:
The landmark trials that established breast conservation therapy (BCT) (breast-conserving surgery followed by adjuvant breast irradiation) as a suitable alternative to mastectomy were conducted in an era that predated biological subtyping of breast cancer and the use of HER2-directed therapies in patients with HER2+ cancers. These trials established adjuvant radiotherapy following breast-conserving surgery as necessary to maximize local control, yet, in the intervening years, overall outcomes have improved significantly owing to widespread adoption of screening mammography, resulting in a substantial reduction in average tumor size at diagnosis, as well as improvements in surgical techniques and, crucial for this proposal, the development of highly active systemic therapies.

Before the development of HER2-targeted therapies, patients with HER2-driven localized breast cancer had among the highest rates of local recurrence. However, with improved identification of these patients and the advent of HER2-directed therapies, outcomes have improved significantly, and trials have sought to optimize treatment to reduce the morbidity of both local and systemic treatment. Among the most salient of these examples is the APT trial, a single-arm adjuvant study that enrolled 410 breast cancer patients with HER2+ tumors ≤ 3cm in size and negative axillary nodes, who received adjuvant systemic therapy with weekly paclitaxel and trastuzumab for 12 weeks (TH) followed by 9 months of trastuzumab monotherapy. In addition to demonstrating a very low incidence of distant recurrence, among those on the trial who underwent BCT (lumpectomy and radiation, n = 244), only 2 local recurrence (LR) events have been reported after 7 years of follow-up (7-year LR = 1.2%), representing among the most favorable local outcomes of any breast cancer cohort studied to date. Confirmatory results are forthcoming from the ATEMPT trial, which evaluated the antibody-drug conjugate T-DM1 (ado-trastuzumab emtansine) (n=383) vs the TH regimen from the APT trial (n = 114), thus far showing only 3 LRs in each arm with a median 3-years of follow-up. Importantly, per the current standard of care for HER2+ patients undergoing BCT, all patients presumably received adjuvant breast radiotherapy.

The balance of the BCT literature, including a landmark meta-analysis by the Early Breast Cancer Trialists' Collaborative Group, suggests that adjuvant radiotherapy approximately halves the risk of local recurrence following lumpectomy across all analyzable subgroups. While the relative benefit appears constant across subgroups, the absolute benefit of adjuvant radiotherapy varies with the underlying risk. Taking the favorable results of the APT trial (1.2% 7-year LR), if one presumes that omission of radiotherapy yields a doubling or tripling of local recurrence (based on the observed RR of 0.5 - 0.66 for those receiving radiotherapy across the preponderance of historical trials), this population might have manifested a LR rate of 2.4 - 3.6% with the omission of radiotherapy. That is to say, the hypothesis is that administration of RT to APT patients undergoing BCT may have reduced the 7-year absolute risk of LR by only 1.2-2.4%. Through the identification of patients who are at low risk of LR, it may be acceptable for such patients to forego radiation. This hypothesis will be studied by evaluating omission of radiotherapy among patients with pT1N0 disease at breast-conserving surgery who receive adjuvant HER2-directed therapy (trastuzumab/paclitaxel preferred, other options per protocol), or with clinical tumors ≤ 3 cm and clinically negative axillary nodes (cN0) who achieve a pathologic complete response (pCR; ypT0N0) following preoperative (neoadjuvant) administration of HER2-directed therapy (trastuzumab/paclitaxel preferred, other options per protocol). It is expcted that the 5-year LR rate for this population omitting radiotherapy will be 2% or less, and that omission of radiation will not have a measurable impact on regional and distant recurrences or overall survival.

The practice of breast radiation oncology has benefited immensely from practice-changing trials that have refined the application of adjuvant radiotherapy since the early surgical studies determined whole breast radiotherapy to be necessary following lumpectomy. There are now several favorable breast cancer subtypes in which patients routinely forego radiotherapy after trials demonstrating modest benefits in terms of local recurrence and no impact on distant recurrence or survival, such as among small, low grade luminal cancers in older women and "good-risk" DCIS. Therefore, this will study the omission of radiotherapy among a population of HER2+ breast cancer patients who are now appreciated to also have favorable risk, so as to similarly weigh the attendant inconveniences, cost and morbidity of radiotherapy in light of an established absolute benefit, which may prove to be modest.

ELIGIBILITY:
Inclusion Criteria:

* The patient or a legally authorized representative must provide study-specific informed consent prior to study entry and, for patients treated in the U.S., authorization permitting release of personal health information.
* female and male patients who have undergone breast conserving surgery and completed a minimum of 4 cycles (12 weeks) of neoadjuvant or adjuvant chemotherapy in combination with HER2-targeted therapy.

  -≥ 40 years of age
* ECOG performance status of 0 ,1, or 2/Karnofsky performance status above 60
* Histologically or cytologically confirmed invasive breast carcinoma.
* tumor must have been determined to be HER2-positive by current ASCO/CAP guidelines based on local testing results.
* Patient must have undergone axillary staging, either sentinel node biopsy (SNB) or axillary lymph nodal dissection (ALND). In neoadjuvant patients, SNB following neoadjuvant therapy is strongly recommended. SNB prior to neoadjuvant therapy is discouraged, but patients are permitted if node negative (pN0).
* The following staging criteria must be met according to AJCC 8th edition criteria:

Adjuvant cohort : By pathologic evaluation, the patient's primary tumor must be </= 2 cm and ipsilateral nodes must be pN0. Surgical lumpectomy margins must be negative for invasive cancer and ductal carcinoma in situ (no ink on tumor).

Neoadjuvant cohort: Prior to neoadjuvant therapy, the patient's primary tumor must be < 3 cm by imaging studies, with negative axillary nodes (cN0) based on axillary U/S, CT, PET or MRI. Physical examination is not sufficient documentation of cN0 status; • Must be ypT0N0 at surgery (lumpectomy); patients with residual non-invasive disease (DCIS) in the surgical specimen (ypTis), are NOT eligible.

* For the Adjuvant cohort, adjuvant therapy must have consisted of a minimum of 4 cycles (12 weeks) of chemotherapy in combination with HER2-targeted therapy.
* For the Neoadjuvant cohort, neoadjuvant therapy must have consisted of a minimum of 4 cycles (12 weeks) of chemotherapy in combination with HER2-targeted therapy.- ; Patients who did not receive chemotherapy in the neoadjuvant setting are not eligible, even if they achieved pCR with their preoperative treatment; nor would these patients become eligible by receiving chemotherapy after surgery.
* In patients assigned to radiation therapy, treatment should start ≤ 12 weeks from surgery on the Neoadjuvant cohort and ≤ 8 weeks from the completion of chemotherapy on the Adjuvant cohort. Patients should continue HER2-targeted therapy during assigned study treatment (radiation or observation).
* Bilateral mammogram or MRI within 52 weeks prior to randomization.
* HIV-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months of randomization are eligible for this trial.

Exclusion Criteria:

* Definitive clinical or radiologic evidence of metastatic disease.
* On the Adjuvant cohort, patients with a primary tumor >2 cm on pathologic examination of the surgical specimen. On the Neoadjuvant cohort, patients with a primary tumor > 3 cm or with abnormal or suspicious ipsilateral axillary nodes by pretreatment imaging, unless demonstrated to be negative by cytologic or histologic examination.
* Pathologically positive axillary nodes at any time including of pN0(i+) or pN0(mol+) ypN0(i+) or ypN0(mol+) disease.
* Patient planning for or status-post mastectomy.
* Radiographically suspicious ipsilateral or contralateral axillary, supraclavicular, infraclavicular, or internal mammary lymph nodes, unless there is histological confirmation that these nodes are negative for metastatic disease.
* Suspicious microcalcifications, densities, or palpable abnormalities (in the ipsilateral or contralateral breast), or mass or non-mass enhancement on MRI (if performed) aside from the known cancer, unless biopsied and found to be benign.
* Non-epithelial breast malignancies such as sarcoma or lymphoma.
* Multicentric carcinoma (invasive cancer or DCIS) in more than one quadrant or separated by > 4 centimeters. If multifocal, all foci should be confined to a maximum tumor bed of 3 cm determined by pathological assessment.
* Paget's disease of the nipple.
* Synchronous (unilateral or bilateral) invasive breast cancer or DCIS. (Patients with synchronous and/or previous contralateral LCIS are eligible.)
* On the Adjuvant cohort, surgical margins that cannot be microscopically assessed or are positive at pathologic evaluation. (If surgical margins are rendered free of disease by re-excision, the patient is eligible).
* Treatment plan that includes regional nodal irradiation.
* Patients treated for a prior invasive breast malignancy are excluded. Contralateral DCIS ≥ 10 years prior to enrollment is permissible.
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.
* Patients on oral, transdermal, or subdermal estrogen replacement (including all estrogen only and estrogen-progesterone formulas) are not eligible unless discontinued prior to randomization.
* Prior ipsilateral breast or thoracic RT for any condition (contralateral RT for DCIS ≥ 10 years prior to randomization is permitted).
* Active collagen vascular disease, specifically dermatomyositis with a CPK level above normal or with an active systemic lupus erythematosus, or scleroderma.
* Clinicians should consider whether any conditions would make this protocol unreasonably hazardous for the patient.
* Pregnancy or lactation at the time of randomization or intention to become pregnant during treatment. (Note: Pregnancy testing according to institutional standards for patients of childbearing potential must be performed within 14 days prior to randomization.)
* Use of any investigational product within 30 days prior to randomization.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1300 (Estimated)
Dates: Start 2023-03-13 (Actual); Primary Completion 2034-02-01 (Estimated); Study Completion 2037-02-01 (Estimated)

PRIMARY OUTCOMES:
recurrence-free interval (RFI) | From randomization to first recurrence event or censoring for the duration of the trial, at 10.5 years
  Time to recurrence event or censoring

SECONDARY OUTCOMES:
ipsilateral breast recurrence (IBR) for radiation omitting arm | From randomization to first recurrence event or censoring for the duration of the trial , measured at year 7
  Time to IBTR event or censoring
ipsilateral breast recurrence (IBR) by treatment arm | From randomization to first recurrence event or censoring for the duration of the trial at 10.5 years.
  Time to ipsilateral breast recurrence (IBR) by treatment arm.
local regional recurrence (LRR) by treatment arm | From randomization to first recurrence event or censoring for the duration of the trial at 10.5 years.
  Time to local regional recurrence (LRR) by treatment arm.
disease-free survival (DFS) by treatment arm. | From the time of randomization for the duration of the trial at 10.5 years.
  To determine disease-free survival (DFS) by treatment arm.
overall survival (OS) by treatment arm. | From the time of randomization for the duration of the trial at 10.5 years.
  To determine overall survival (OS) by treatment arm.
patient-reported breast pain by treatment arm using the Breast Cancer Treatment Outcome Scale (BCTOS) | At 3 years after randomization
  To evaluate whether there is a difference in patient-reported breast pain in patients who do and do not receive breast radiation in cohort A and cohort B. The BCTOS pain score has a range from 1-5 with higher scores indicating worse pain.
patient-reported worry about recurrence by treatment arm using a the three-item worry about recurrence score | At 3 years after randomization
  To evaluate whether there is a difference in patient-reported worry about recurrence in patients who do and do not receive breast radiation in cohort A and cohort B. The worry about recurrence score has a range from 1-5 with higher scores indicating more worry.

CONTACTS AND LOCATIONS:
Overall Officials: Norman Wolmark, MD, Principal Investigator — NRG Oncology
Locations (416):
- United States (411):
  - Cancer Center at Saint Joseph's, Phoenix, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - University of Arizona Cancer Center-North Campus, Tucson, Arizona
  - NEA Baptist Memorial Hospital and Fowler Family Cancer Center - Jonesboro, Jonesboro, Arkansas
  - Kaiser Permanente-Deer Valley Medical Center, Antioch, California
  - Mission Hope Medical Oncology - Arroyo Grande, Arroyo Grande, California
  - PCR Oncology, Arroyo Grande, California
  - Sutter Auburn Faith Hospital, Auburn, California
  - Sutter Cancer Centers Radiation Oncology Services-Auburn, Auburn, California
  - Tower Cancer Research Foundation, Beverly Hills, California
  - Sutter Cancer Centers Radiation Oncology Services-Cameron Park, Cameron Park, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Kaiser Permanente Dublin, Dublin, California
  - Kaiser Permanente-Fremont, Fremont, California
  - Palo Alto Medical Foundation-Fremont, Fremont, California
  - Fresno Cancer Center, Fresno, California
  - Kaiser Permanente-Fresno, Fresno, California
  - UCI Health - Chao Family Comprehensive Cancer Center and Ambulatory Care, Irvine, California
  - City of Hope at Irvine Lennar, Irvine, California
  - City of Hope Antelope Valley, Lancaster, California
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Memorial Medical Center, Modesto, California
  - Kaiser Permanente-Modesto, Modesto, California
  - Palo Alto Medical Foundation-Camino Division, Mountain View, California
  - Kaiser Permanente Oakland-Broadway, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Palo Alto Medical Foundation Health Care, Palo Alto, California
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - Pomona Valley Hospital Medical Center, Pomona, California
  - Kaiser Permanente-Rancho Cordova Cancer Center, Rancho Cordova, California
  - Kaiser Permanente- Marshall Medical Offices, Redwood City, California
  - Kaiser Permanente-Richmond, Richmond, California
  - Rohnert Park Cancer Center, Rohnert Park, California
  - Kaiser Permanente-Roseville, Roseville, California
  - Sutter Cancer Centers Radiation Oncology Services-Roseville, Roseville, California
  - Sutter Roseville Medical Center, Roseville, California
  - The Permanente Medical Group-Roseville Radiation Oncology, Roseville, California
  - Kaiser Permanente Downtown Commons, Sacramento, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Kaiser Permanente-South Sacramento, Sacramento, California
  - South Sacramento Cancer Center, Sacramento, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Stanford Cancer Center South Bay, San Jose, California
  - Kaiser Permanente San Leandro, San Leandro, California
  - Pacific Central Coast Health Center-San Luis Obispo, San Luis Obispo, California
  - Kaiser San Rafael-Gallinas, San Rafael, California
  - Ridley-Tree Cancer Center, Santa Barbara, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Mission Hope Medical Oncology - Santa Maria, Santa Maria, California
  - Kaiser Permanente-Santa Rosa, Santa Rosa, California
  - Sutter Pacific Medical Foundation, Santa Rosa, California
  - City of Hope South Pasadena, South Pasadena, California
  - Kaiser Permanente Cancer Treatment Center, South San Francisco, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Kaiser Permanente-Stockton, Stockton, California
  - Palo Alto Medical Foundation-Sunnyvale, Sunnyvale, California
  - Cedars-Sinai Cancer - Tarzana, Tarzana, California
  - City of Hope South Bay, Torrance, California
  - Torrance Memorial Physician Network - Cancer Care, Torrance, California
  - City of Hope Upland, Upland, California
  - Kaiser Permanente Medical Center-Vacaville, Vacaville, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - UCHealth Memorial Hospital Central, Colorado Springs, Colorado
  - Memorial Hospital North, Colorado Springs, Colorado
  - Saint Francis Cancer Center, Colorado Springs, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Cancer Care and Hematology-Fort Collins, Fort Collins, Colorado
  - UCHealth Greeley Hospital, Greeley, Colorado
  - UCHealth Highlands Ranch Hospital, Highlands Ranch, Colorado
  - Medical Center of the Rockies, Loveland, Colorado
  - John Fitzgerald Kennedy Medical Center, Atlantis, Florida
  - Morton Plant Hospital, Clearwater, Florida
  - Lee Memorial Health System, Fort Myers, Florida
  - Regional Cancer Center-Lee Memorial Health System, Fort Myers, Florida
  - Sarasota Memorial Hospital-Venice, N. Venice, Florida
  - Health Central, Ocoee, Florida
  - Orlando Health Cancer Institute, Orlando, Florida
  - GenesisCare USA - Plantation, Plantation, Florida
  - Florida Cancer Specialists - Sarasota, Sarasota, Florida
  - Intercoastal Medical Group - Cattleridge II, Sarasota, Florida
  - Florida Cancer Specialists - Sarasota Downtown, Sarasota, Florida
  - First Physicians Group - Urology Robotic and Minimally Invasive Surgery, Sarasota, Florida
  - First Physicians Group-Sarasota, Sarasota, Florida
  - Sarasota Memorial Hospital, Sarasota, Florida
  - Sarasota Memorial Health Care Center at University Parkway, Sarasota, Florida
  - Moffitt Cancer Center-International Plaza, Tampa, Florida
  - Moffitt Cancer Center - McKinley Campus, Tampa, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Florida Cancer Specialists - Venice Pinebrook, Venice, Florida
  - Florida Cancer Specialists - Venice Island, Venice, Florida
  - Moffitt Cancer Center at Wesley Chapel, Wesley Chapel, Florida
  - Grady Health System, Atlanta, Georgia
  - Emory Proton Therapy Center, Atlanta, Georgia
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Emory Decatur Hospital, Decatur, Georgia
  - Emory Johns Creek Hospital, Johns Creek, Georgia
  - CTCA at Southeastern Regional Medical Center, Newnan, Georgia
  - South Georgia Medical Center/Pearlman Cancer Center, Valdosta, Georgia
  - Hawaii Cancer Care Inc - Waterfront Plaza, Honolulu, Hawaii
  - Queen's Cancer Cenrer - POB I, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Kuakini Medical Center, Honolulu, Hawaii
  - Queen's Cancer Center - Kuakini, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Castle Medical Center, Kailua, Hawaii
  - Wilcox Memorial Hospital and Kauai Medical Clinic, Lihue, Hawaii
  - Hawaii Cancer Care - Westridge, ‘Aiea, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Queen's Cancer Center - Pearlridge, ‘Aiea, Hawaii
  - The Cancer Center of Hawaii-Pali Momi, ‘Aiea, Hawaii
  - The Queen's Medical Center - West Oahu, ‘Ewa Beach, Hawaii
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - Rush-Copley Medical Center, Aurora, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Saint Mary's Hospital, Centralia, Illinois
  - Northwestern University, Chicago, Illinois
  - John H Stroger Jr Hospital of Cook County, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Northwestern Medicine Cancer Center Kishwaukee, DeKalb, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Elmhurst Memorial Hospital, Elmhurst, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - Northwestern Medicine Glenview Outpatient Center, Glenview, Illinois
  - Northwestern Medicine Grayslake Outpatient Center, Grayslake, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Northwestern Medicine Lake Forest Hospital, Lake Forest, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Edward Hospital/Cancer Center, Naperville, Illinois
  - UC Comprehensive Cancer Center at Silver Cross, New Lenox, Illinois
  - Carle Cancer Institute Normal, Normal, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - HSHS Saint Elizabeth's Hospital, O'Fallon, Illinois
  - Northwestern Medicine Orland Park, Orland Park, Illinois
  - University of Chicago Medicine-Orland Park, Orland Park, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Midwestern Regional Medical Center, Zion, Illinois
  - Northwest Cancer Center - Main Campus, Crown Point, Indiana
  - UChicago Medicine Northwest Indiana, Crown Point, Indiana
  - Northwest Oncology LLC, Dyer, Indiana
  - Goshen Center for Cancer Care, Goshen, Indiana
  - Northwest Cancer Center - Hobart, Hobart, Indiana
  - Saint Mary Medical Center, Hobart, Indiana
  - The Community Hospital, Munster, Indiana
  - Women's Diagnostic Center - Munster, Munster, Indiana
  - Reid Health, Richmond, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Northwest Cancer Center - Valparaiso, Valparaiso, Indiana
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic - Ames, Ames, Iowa
  - UI Health Care Mission Cancer and Blood - Ankeny Clinic, Ankeny, Iowa
  - Physicians' Clinic of Iowa PC, Cedar Rapids, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - UI Health Care Mission Cancer and Blood - West Des Moines Clinic, Clive, Iowa
  - Greater Regional Medical Center, Creston, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Des Moines Clinic, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Laurel Clinic, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Waukee Clinic, Waukee, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - University of Kansas Cancer Center, Kansas City, Kansas
  - The University of Kansas Cancer Center - Olathe, Olathe, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - University of Kansas Hospital-Indian Creek Campus, Overland Park, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - University of Kansas Health System Saint Francis Campus, Topeka, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - The James Graham Brown Cancer Center at University of Louisville, Louisville, Kentucky
  - UofL Health Medical Center Northeast, Louisville, Kentucky
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - UM Upper Chesapeake Medical Center, Bel Air, Maryland
  - Central Maryland Radiation Oncology in Howard County, Columbia, Maryland
  - University of Maryland Shore Medical Center at Easton, Easton, Maryland
  - UM Baltimore Washington Medical Center/Tate Cancer Center, Glen Burnie, Maryland
  - UM Capital Region Medical Center, Largo, Maryland
  - Bronson Battle Creek, Battle Creek, Michigan
  - Henry Ford Cancer Institute-Downriver, Brownstown, Michigan
  - Caro Cancer Center, Caro, Michigan
  - Michigan Healthcare Professionals Clarkston, Clarkston, Michigan
  - Henry Ford Macomb Hospital-Clinton Township, Clinton Township, Michigan
  - Henry Ford Medical Center-Fairlane, Dearborn, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - OSF Saint Francis Hospital and Medical Group, Escanaba, Michigan
  - Michigan Healthcare Professionals Farmington, Farmington Hills, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - Corewell Health Grand Rapids Hospitals - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Trinity Health Grand Rapids Hospital, Grand Rapids, Michigan
  - Allegiance Health, Jackson, Michigan
  - Michigan Healthcare Professionals Macomb, Macomb, Michigan
  - Michigan Healthcare Professionals Madison Heights, Madison Heights, Michigan
  - Saint Mary's Oncology/Hematology Associates of Marlette, Marlette, Michigan
  - Henry Ford Medical Center-Columbus, Novi, Michigan
  - Trinity Health Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - Corewell Health William Beaumont University Hospital, Royal Oak, Michigan
  - MyMichigan Medical Center Saginaw, Saginaw, Michigan
  - Oncology Hematology Associates of Saginaw Valley PC, Saginaw, Michigan
  - MyMichigan Medical Center Tawas, Tawas City, Michigan
  - Corewell Health Beaumont Troy Hospital, Troy, Michigan
  - Michigan Healthcare Professionals Troy, Troy, Michigan
  - Henry Ford West Bloomfield Hospital, West Bloomfield, Michigan
  - Saint Mary's Oncology/Hematology Associates of West Branch, West Branch, Michigan
  - University of Michigan Health - West, Wyoming, Michigan
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Essentia Health Saint Joseph's Medical Center, Brainerd, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health - Deer River Clinic, Deer River, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Saint Mary's Medical Center, Duluth, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Saint Luke's Hospital of Duluth, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Essentia Health Hibbing Clinic, Hibbing, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Monticello Cancer Center, Monticello, Minnesota
  - Coborn Cancer Center at Saint Cloud Hospital, Saint Cloud, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Essentia Health Sandstone, Sandstone, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Essentia Health Virginia Clinic, Virginia, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Baptist Memorial Hospital and Cancer Center-Golden Triangle, Columbus, Mississippi
  - Baptist Cancer Center-Grenada, Grenada, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Union County, New Albany, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Oxford, Oxford, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Desoto, Southhaven, Mississippi
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Parkland Health Center - Farmington, Farmington, Missouri
  - University of Kansas Cancer Center - North, Kansas City, Missouri
  - University of Kansas Cancer Center - Lee's Summit, Lee's Summit, Missouri
  - University of Kansas Cancer Center at North Kansas City Hospital, North Kansas City, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - BJC Outpatient Center at Sunset Hills, Sunset Hills, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Nebraska Medicine-Bellevue, Bellevue, Nebraska
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Cancer Partners of Nebraska, Lincoln, Nebraska
  - Nebraska Medicine-Village Pointe, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - OptumCare Cancer Care at Seven Hills, Henderson, Nevada
  - OptumCare Cancer Care at Charleston, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Central, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Southeast, Las Vegas, Nevada
  - OptumCare Cancer Care at MountainView, Las Vegas, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Northwell Health Imbert Cancer Center, Bay Shore, New York
  - Sands Cancer Center, Canandaigua, New York
  - Memorial Sloan Kettering Commack, Commack, New York
  - Noyes Memorial Hospital/Myers Cancer Center, Dansville, New York
  - Northwell Health Cancer Institute at Huntington, Greenlawn, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Northwell Health/Center for Advanced Medicine, Lake Success, New York
  - Northern Westchester Hospital, Mount Kisco, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Upstate Cancer Center at Oswego, Oswego, New York
  - Wilmot Cancer Institute Radiation Oncology at Greece, Rochester, New York
  - Highland Hospital, Rochester, New York
  - Pluta Cancer Center, Rochester, New York
  - University of Rochester, Rochester, New York
  - Phelps Memorial Hospital Center, Sleepy Hollow, New York
  - Staten Island University Hospital, Staten Island, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - SUNY Upstate Medical Center-Community Campus, Syracuse, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Montefiore Medical Center-Weiler Hospital, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
  - Upstate Cancer Center at Verona, Verona, New York
  - Wilmot Cancer Institute at Webster, Webster, New York
  - East Carolina University, Greenville, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Indu and Raj Soin Medical Center, Beavercreek, Ohio
  - Cleveland Clinic Mercy Hospital, Canton, Ohio
  - Dayton Physicians LLC-Miami Valley South, Centerville, Ohio
  - Miami Valley Hospital South, Centerville, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Premier Blood and Cancer Center, Dayton, Ohio
  - Dayton Physician LLC - Englewood, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Dublin Methodist Hospital, Dublin, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Dayton Physicians LLC-Atrium, Franklin, Ohio
  - Miami Valley Cancer Care and Infusion, Greenville, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - OhioHealth Mansfield Hospital, Mansfield, Ohio
  - OhioHealth Marion General Hospital, Marion, Ohio
  - Dayton Physicians LLC - Troy, Troy, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Saint Charles Health System, Bend, Oregon
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Cancer Institute Clackamas Clinic, Clackamas, Oregon
  - Legacy Mount Hood Medical Center, Gresham, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Legacy Good Samaritan Hospital and Medical Center, Portland, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Legacy Meridian Park Hospital, Tualatin, Oregon
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - UPMC-Magee Womens Hospital, Pittsburgh, Pennsylvania
  - Women and Infants Hospital, Providence, Rhode Island
  - Kent Hospital, Warwick, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Lexington Medical Center, West Columbia, South Carolina
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Baptist Memorial Hospital and Cancer Center-Collierville, Collierville, Tennessee
  - Baptist Memorial Hospital and Cancer Center-Memphis, Memphis, Tennessee
  - MD Anderson in The Woodlands, Conroe, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - MD Anderson West Houston, Houston, Texas
  - MD Anderson League City, League City, Texas
  - MD Anderson in Sugar Land, Sugar Land, Texas
  - Farmington Health Center, Farmington, Utah
  - University of Utah Sugarhouse Health Center, Salt Lake City, Utah
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - University of Vermont Medical Center, Burlington, Vermont
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - Dartmouth Cancer Center - North, Saint Johnsbury, Vermont
  - Bon Secours Memorial Regional Medical Center, Mechanicsville, Virginia
  - Bon Secours Saint Francis Medical Center, Midlothian, Virginia
  - Bon Secours Saint Mary's Hospital, Richmond, Virginia
  - Bon Secours Cancer Institute at Reynolds Crossing, Richmond, Virginia
  - Swedish Cancer Institute-Edmonds, Edmonds, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Skagit Regional Health Cancer Care Center, Mount Vernon, Washington
  - Swedish Medical Center-Ballard Campus, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - Legacy Cancer Institute Medical Oncology and Day Treatment, Vancouver, Washington
  - Legacy Salmon Creek Hospital, Vancouver, Washington
  - Langlade Hospital and Cancer Center, Antigo, Wisconsin
  - Duluth Clinic Ashland, Ashland, Wisconsin
  - Northwest Wisconsin Cancer Center, Ashland, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Essentia Health-Hayward Clinic, Hayward, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Froedtert Menomonee Falls Hospital, Menomonee Falls, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - ProHealth D N Greenwald Center, Mukwonago, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - Drexel Town Square Health Center, Oak Creek, Wisconsin
  - ProHealth Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Aspirus Cancer Care - James Beck Cancer Center, Rhinelander, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sheboygan, Sheboygan, Wisconsin
  - Sheboygan Physicians Group, Sheboygan, Wisconsin
  - Essentia Health-Spooner Clinic, Spooner, Wisconsin
  - Aspirus Cancer Care - Stevens Point, Stevens Point, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Essentia Health Saint Mary's Hospital - Superior, Superior, Wisconsin
  - UW Cancer Center at ProHealth Care, Waukesha, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin
  - Froedtert West Bend Hospital/Kraemer Cancer Center, West Bend, Wisconsin
  - Aspirus Cancer Care - Wisconsin Rapids, Wisconsin Rapids, Wisconsin
- Puerto Rico (5):
  - Cancer Center-Metro Medical Center Bayamon, Bayamón
  - Doctors Cancer Center, Manatí
  - San Juan Community Oncology Group, San Juan
  - Centro Comprensivo de Cancer de UPR, San Juan
  - San Juan City Hospital, San Juan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Braunstein LZ, Mitchell MP, Bandos H, Sikov WM, Khan AJ, Chen PY, Ganz PA, Jagsi R, White JR, Cecchini RS, Kang H, Puhalla SL, Bolton KL, Connolly EP, Stringer-Reasor EM, Gergelis KR, Julian TB, Mamounas EP, Wolmark N. NRG-BR008/HERO study: a Phase III randomized trial of radiotherapy optimization for low-risk HER2-positive breast cancer. Future Oncol. 2025 Jul;21(16):2017-2025. doi: 10.1080/14796694.2025.2511586. Epub 2025 Jun 26. PMID 40574381